CLINICAL TRIAL: NCT05292547
Title: Substance Misuse To Psychiatric Disorders-Repetitive Transcranial Magnetic Stimulation to People With Cannabis Use Disorder
Brief Title: Repetitive Transcranial Magnetic Stimulation to People With Cannabis Use Disorder (SToP-C-rTMS x CUD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW21-656
Record Dates: First submitted 2022-03-13; First posted 2022-03-23 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Cannabis Use Disorder; Repetitive Transcranial Magnetic Stimulation
Keywords: Cannabis; TMS
MeSH Terms: conditions — Marijuana Abuse | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Active Comparator): Subjects receive 20 rTMS sessions in 2 weeks
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Arm 2 (Active Comparator): Subjects receive 20 rTMS sessions in 4 weeks
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Arm 3 (Active Comparator): Subjects receive 20 rTMS sessions in 5 weeks
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — rTMS using Magventure TMS system is delivered at the dorsolateral prefrontal cortex of consented subjects according to 3 different stimulation schedules.

SUMMARY:
This study is to explore if repetitive transcrinal magnetic stimulation (rTMS) with different stimulation schedules will be equally effective in reducing carving, frequency of cannabis use, and the severity of cannabis use disorder in participants suffering from cannabis use disorder (CUD).

The investigators assume the hypotheses as:

1. Multiple rTMS sessions can reduce craving for cannabis, severity of CUD, frequency and amount of cannabis use.
2. Different rTMS treatment schedules have differences in reducing the craving for cannabis and severity of CUD, and prolonging relapse of cannabis use.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and communicate in English and/or Chinese SToP-C-rTMS x CUD
* Able to give informed consent
* Using cannabis or marijuana as the primary psychoactive substance of abuse
* Diagnosed with Cannabis Use Disorder according to the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) by the Structured Clinical Interview for DSM-5 Disorders (SCID-5)

Exclusion Criteria:

* Age <18 years old
* Unable to read English or Chinese
* Unable to give informed consent
* Had been diagnosed with the following disorders, including neurodevelopmental disorders, DSM-5 defined substance use disorder greater than moderate in severity, and neurocognitive disorders
* Contra-indicated to have rTMS, including subjects with electronic and/or magnetic implants (e.g. pacemaker, implantable cardioverter defibrillator [ICD], cerebral shunts, cochlear implant, etc.), with metallic or mechanic fragments (e.g., screws, plates, stents, clips, etc.), pregnant, with any known or history of neurological conditions including cerebral vascular accidents, epilepsy, brain tumor or space occupying lesion, poorly controlled or unstable diabetes mellitus, and receiving unstable dose(s) of antipsychotics, antidepressants, benzodiazepines and/or anticonvulsants in the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
A change in amount of cannabis use | 12 months
  Subject's self-report on the amount of cannabis use (in terms of number of joints per day) at baseline to the amount of use at 2nd week, 4th week, 5th week, 3rd month, 6th month and 12-month post-treatment with rTMS
A change in frequency of Cannabis Use | 12 months
  Subject's self-repot on the frequency of cannabis use (in terms of number of times of use per day and/or per week) at baseline to that at 2nd week, 4th week, 5th week, 3rd month, 6th month and 12-month post-treatment with rTMS
Severity of Cannabis Use Disorder | 12 months
  A change in severity of cannabis use disorder measured by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) with severity ranges from 0 to 11 (maximum severity) from baseline to that at 2nd week, 4th week, 5th week, 3rd month, 6th month and 12-month post-treatment with rTMS
Severity of Dependence | 12 months
  A change in scorings measured by the Severity of Dependence Scale (ranges from a minimum of 5 to a maximum of 20) from baseline to that at 2nd week, 4th week, 5th week, 3rd month, 6th month and 12-month post-treatment with rTMS
Craving | 12 months
  A change in scorings measured by Marijuana Craving Questionnaire (ranges from a minimum of 17 to a maximum of 119) from baseline to to that at 2nd week, 4th week, 5th week, 3rd month, 6th month and 12-month post-treatment with rTMS

SECONDARY OUTCOMES:
Level of Anxiety | 12 months
  A change in severity of anxiety measured by Beck Anxiety Inventory (with a score from a minimum of 0 to a maximum of 63) at baseline to that at 2nd week, 4th week, 5th week, 3rd month, 6th month and 12-month post-treatment with rTMS
Level of Depression | 12 months
  A change in severity of depression measured by Beck Depression Inventory (with a score from a minimum of 0 to a maximum of 63) at baseline to that at at 2nd week, 4th week, 5th week, 3rd month, 6th month and 12-month post-treatment with rTMS

CONTACTS AND LOCATIONS:
Overall Officials: Albert KK Chung, MBBS, Principal Investigator — Department of Psychiatry, The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong